CLINICAL TRIAL: NCT03562650
Title: Computerized Treatment for Social Anxiety
Brief Title: Text Message Treatment for Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017.22461
Record Dates: First submitted 2018-02-05; First posted 2018-06-19 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Social Anxiety

STUDY DESIGN:
Intervention Model Description: Active treatment and active treatment control conditions.
Who Masked: Participant
Masking Description: All participants are assigned to a condition and given a treatment justification, but are not told whether they are in the treatment or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Behavior Fading (Experimental): Participants are asked to pick their three most common safety behaviors from a list and then receive texts every other day for a month reminding them to fade those behaviors.
  Interventions: Behavioral: Safety Behavior Fading
- Present Centered (Active Comparator): Participants receive texts every other day for a month asking them to try to focus on the present that day.
  Interventions: Behavioral: Present Centered

INTERVENTIONS:
Behavioral: Safety Behavior Fading — Participants are asked to fade their three most common safety behaviors associated with their social anxiety
  Arms: Safety Behavior Fading
Behavioral: Present Centered — Participants are asked to try to increase their focus on the present.
  Arms: Present Centered

SUMMARY:
This is an intervention study designed to evaluate a text message based safety behavior fading treatment for people with social anxiety disorder.

DETAILED DESCRIPTION:
This study hopes to assess whether a month long text message based safety behavior fading protocol is effective in reducing safety behaviors and social anxiety symptoms. Over the course of four consecutive weeks, text messages will be sent to participants the first day of the study and every other day for four weeks (14 texts in total). These text messages will remind participants to either avoid using their three most engaged in safety behaviors (assessed at pre-treatment) or to stay present-focused. The past week frequency of the participants' safety behaviors will be assessed at the beginning of pre-treatment, post-treatment, and four week follow up assessments Participants will be asked to complete an additional online questionnaire for both a post-treatment and a 4-week post-treatment follow up assessment. We hypothesize that: 1) the safety behavior group will show a greater overall reduction in social anxiety symptoms, 2) that the safety behavior group will show a reduction in the frequency of safety behavior use, and 3) that the present-focused group will show an increase in mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* Social Phobia Inventory score > 29

Exclusion Criteria:

* receiving therapy
* changes in the past 4 weeks with medication for emotional difficulties
* psychotic symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-01-27 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Social Phobia Inventory (SPIN) | Change in social anxiety symptoms from baseline to post treatment (4 weeks) and one month follow up (8 weeks)
  Self-report scale that measures Social anxiety symptoms. Scores range from 0 to 68 with higher scores indicating higher levels of social anxiety symptoms.

SECONDARY OUTCOMES:
Subtle Avoidance Frequency Examination(SAFE) | Change in safety behavior use from baseline to post treatment (4 weeks) and one month follow up (8 weeks)
  Self report scale used to assess how often people use safety behaviors to cope with their anxiety. Scores range from 33 to 165. Higher total scores are associated with more frequent safety behavior use.
Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | Change in mindfulness from baseline to post treatment (4 weeks) and one month follow up (8 weeks)
  Self-report used to measure mindfulness, including awareness of thoughts and feelings. Total scores range from 12 to 48 with higher scores indicating a greater ability to be mindful, present in the moment, and aware of thoughts and feelings.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Department of Psychology, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cougle JR, Mueller NE, McDermott KA, Wilver NL, Carlton CN, Okey SA. Text message safety behavior reduction for social anxiety: A randomized controlled trial. J Consult Clin Psychol. 2020 May;88(5):445-454. doi: 10.1037/ccp0000494. Epub 2020 Feb 27. PMID 32105093